CLINICAL TRIAL: NCT07139171
Title: Study on the Role and Mechanism of Plasma Exosome microRNAs in Cognitive Impairment in First-episode Schizophrenia
Status: Recruiting | Type: Observational
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FESW-TJAH
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia; cognitive funciton; exosome; microRNA
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Schizophrenic Patients: 200 individuals aged 18-65 years meeting DSM-5 criteria for schizophrenia or schizophreniform disorder. Participants must be in their first illness episode and either completely antipsychotic-naïve or have received antipsychotic medication for ≤ 4 weeks lifetime and ≤ 2 weeks immediately before enrollment. All provide written informed consent.
- Healthy Control: 100 Han Chinese volunteers aged 18-65 years who are group-matched to patients on sex, age, and education. All have no personal history of any psychiatric disorder, no family history of psychotic illness in first- or second-degree relatives and provide written informed consent.

SUMMARY:
Schizophrenia is a severe mental illness characterised by positive symptoms, negative symptoms, and cognitive symptoms. In recent years, an increasing number of doctors and scholars have focused on cognitive symptoms; however, the mechanisms underlying cognitive impairment remain unclear. Recently, exosome research methods have provided new avenues for investigation. This study applies exosome research methods to first-episode, drug-naive schizophrenia patients to explore gene expression changes associated with cognitive impairment and gain a deeper understanding of the mechanisms underlying cognitive impairment. By integrating basic research with clinical findings, we aim to further investigate the molecular mechanisms underlying cognitive impairment in schizophrenia patients, identify potential intervention targets, and provide insights for future drug development.

DETAILED DESCRIPTION:
This single-center, prospective cohort study will enroll 200 drug-naive schizophrenia patients and 100 demographically matched healthy volunteers to identify biological signatures of cognitive impairment and to develop predictive models for subsequent change. At baseline we will administer the MATRICS Consensus Cognitive Battery (MCCB), clinical rating scales, multimodal magnetic resonance imaging (MRI), and collect fasting blood and first-morning urine for multi-omics assays. Participants are re-evaluated at 4, 8 and 12 weeks during naturalistic antipsychotic treatment, repeating cognitive testing, clinical scales, and blood/urine sampling. Primary analyses will link baseline omics to the MCCB overall composite score; secondary analyses will model the longitudinal trajectories of both cognition and biomarkers to derive parsimonious predictors of cognitive gain versus persistent impairment. The resulting biomarker panels are expected to inform future stratified clinical trials and mechanism-based cognitive remediation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers matched to the patient group on sex, age, and education level;
* No family history of psychiatric disorders among first- or second-degree relatives (two generations);
* Ethnic Han Chinese;
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Any serious physical illness, including but not limited to uncontrolled hypertension, severe cardiovascular, cerebrovascular, pulmonary, thyroid, or metabolic disease, diabetes, epilepsy, or metabolic syndrome;
* Current or past diagnosis of substance-induced psychotic disorder, delusional disorder, brief psychotic disorder, or mood disorder with psychotic features;
* Pregnancy or breastfeeding;
* Any condition that would interfere with the ability to give informed consent or complete study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will recruit two groups from the outpatient and inpatient services of Tianjin Anding Hospital and surrounding communities in Tianjin, China. The patient cohort will consist of 200 Han Chinese adults aged 18-65 years who are in their first episode of schizophrenia or schizophreniform disorder and have never received antipsychotics or received them for ≤4 weeks lifetime and ≤2 weeks immediately before enrollment. The healthy control cohort will include 100 Han Chinese adults matched to the patient group on sex, age, and education; they must have no personal or family history of major psychiatric disorders and show no cognitive impairment on formal testing.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | Baseline, week8
  All participants underwent cognitive function assessment based on the MATRICS Consensus Cognitive Battery (MCCB). The battery covers seven cognitive domains and two composite scores. The MCCB scoring procedure generates standardised T-scores that are corrected for age, gender, and educational level. Higher T-scores indicate better cognitive function.
Plasma Exosome Concentration | Baseline
  Fasting plasma samples collected at baseline will be processed by standard ultracentrifugation and nanoparticle tracking analysis (NTA) to quantify total exosome concentration, expressed as particles/mL. This single parameter will serve as the primary biomarker to evaluate its association with cognitive impairment in antipsychotic-naïve schizophrenia patients
The MicroRNA Expression Profile | Baseline
  Levels of microRNAs isolated from plasma-derived exosomes at baseline, quantified by Quantitative Reverse Transcription Polymerase Chain Reaction using a validated panel of schizophrenia- and cognition-related miRNAs, reported as fold-change relative to exogenous spike-in control.
Plasma Exosome Size Distribution | Baseline
  Fasting plasma samples collected at baseline will be processed by standard ultracentrifugation and nanoparticle tracking analysis (NTA) to quantify total exosome size distribution (mode, mean, and particle diameter range), expressed as particles/mL. This single parameter will serve as the primary biomarker to evaluate its association with cognitive impairment in antipsychotic-naïve schizophrenia patients

SECONDARY OUTCOMES:
Psychiatric Symptoms | Baseline, week4, week8, week12
  The psychiatric symptoms of schizophrenia were assessed in all enrolled patients using the Positive and Negative Syndrome Scale (PANSS). The PANSS is a 30-item clinician-rated scale yielding a total score ranging from 30 (least symptomatic) to 210 (symptomatic), where higher scores indicate more severe psychopathology.
Depressive Symptoms | Baseline, week4, week8, week12
  The Hamilton Depression Scale-24 (HAMD-24) was used to assess the severity of depressive symptoms. Each item was scored on a scale of 0 (none) to 4 (severe); the total score ranged from 0 to 76, with higher scores indicating more severe depressive symptoms.
Anxiety Symptoms | baseline, week 4, week 8 and week 12
  The Hamilton Anxiety Scale (HAMA) is used to assess the severity of anxiety symptoms. Each item is scored on a scale of 0 (none) to 4 (very severe), with a total score range of 0-56. Higher scores indicate more severe anxiety symptoms.
Sleep Quality | baseline, week 4, week 8 and week 12
  The Pittsburgh Sleep Quality Index (PSQI) is used to assess sleep quality and sleep disorders over the past month. The questionnaire includes seven subscale scores (subjective sleep quality, sleep onset latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication use, and daytime functioning), with each subscale scored on a scale of 0 to 3. The sum of the seven subscale scores constitutes the PSQI total score, ranging from 0 to 21, with higher scores indicating poorer sleep quality.
Aggressive behaviors | Baseline
  The Modified Open Aggression Scale (MOAS) is a four-component scale administered by clinicians or observers that quantifies verbal aggression, aggression toward objects, self-aggression, and physical aggression toward others. Each component consists of five items, with scores ranging from 0 (none) to 4 (extreme). The scores from each component are added together to produce a total weighted score ranging from 0 to 40, with higher scores indicating more severe overall aggressive behaviour.
Brain Magnetic Resonance Imaging (MRI) | Baseline
  Multimodal 3 T MRI acquired at baseline, including T1-weighted anatomical imaging, diffusion tensor imaging (DTI) and resting-state functional MRI. Extracted metrics-cortical thickness, regional gray-matter volume, fractional anisotropy, mean diffusivity, and amplitude of low-frequency fluctuation-will be used to quantify structural and functional alterations associated with cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, China